CLINICAL TRIAL: NCT06879158
Title: A Randomized, Open-label, Fasting, Single Dose, Two-way Crossover Study to Evaluate the Pharmacokinetics and Safety of BR3409 and Co-administration of BR3409-1 and BR3409-2 in Healthy Volunteers
Brief Title: A Study to Evaluate the Pharmacokinetics and Safety of BR3409 and Co-administration of BR3409-1 and BR3409-2 in Healthy Volunteers Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-ELMC-CT-101
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BR3409 (Experimental)
  Interventions: Drug: BR3409
- BR3409-1 + BR3409-2 (Active Comparator)
  Interventions: Drug: BR3409-1; Drug: BR3409-2

INTERVENTIONS:
Drug: BR3409 — One tablet administered alone
  Arms: BR3409
Drug: BR3409-1 — One tablet administered alone
  Arms: BR3409-1 + BR3409-2
Drug: BR3409-2 — One tablet administered alone
  Arms: BR3409-1 + BR3409-2

SUMMARY:
The purpose of this clinical study is to evaluate the pharmacokinetics and safety of BR3409 and co-administration of BR3409-1 and BR3409-2 in healthy volunteers Under Fasting Conditions

ELIGIBILITY:
Inclusion Criteria:

* Those have body mass index (BMI: weight(kg)/the square of {height(m)}) within the range of 18.0 to 30.0 at screening visit.

  * For men, Those who weigh 55 kg or more
  * For women, Those who weigh 50 kg or more
* Those who sign written consent spontaneously after listening to and understanding sufficient explanation of the purpose and contents of this clinical trial, characteristics of the Investigational products, expected adverse events, etc.
* Those who agree to rule out the possibility of their and their spouses' or sexual partners' pregnancy by using methods of contraception accepted in clinical trial*(Except for hormone drugs) from the date of consent to 56 days after the last administration and disagree to provide their sperm or ovum.

  * Methods of contraception accepted in clinical trial: Combined use of intrauterine device, vasectomy, tubal ligation, and barrier methods (male condom, female condom, cervical cap, contraceptive diaphragm, sponge, etc.) or combined use of two or more barrier methods if spermicide is used.

Exclusion Criteria:

* Those who have taken drugs that induce and inhibit metabolizing enzymes such as barbiturate within 30 days before the first administration date or have taken drugs concerned about affecting this clinical trial within 10 days before the first administration date. (However, participation is possible considering pharmacokinetics and pharmacodynamics such as Interaction of investigational products, half-life of concomitant drugs, etc.)
* Those who have participated in other clinical trials(including bioequivalence tests) and administered their investigational products within 6 months before the first day of administration. (However, the termination for participation in other clinical trials are based on the last administration date of their investigational products)
* Those who have a medical history of gastrointestinal resection or gastrointestinal diseases that may affect the absorption of drugs. (Except for simple appendectomy, hernia surgery)
* In the case of a female subject, those suspected pregnancy or pregnant woman, lactating woman.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-11-10 (Actual); Primary Completion 2025-01-26 (Actual); Study Completion 2025-01-26 (Actual)

PRIMARY OUTCOMES:
AUCτ | 0~72 hours after administration
  Area under the plasma drug concentration-time curve from 0 to time τ
Cmax | 0~72 hours after administration
  Maximum Concentration of Drug in Plasma

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center, H PLUS Yangji Hospital, Seoul, Gwanakgu, South Korea

IPD SHARING:
Plan to Share IPD: No